CLINICAL TRIAL: NCT07316101
Title: Clinical Trial of an Anti-Fog Drainage Device for Endoscopic Endonasal Sellar Region Tumor Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WestChinaH-HX-2025-06
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Pituitary Adenoma; Craniopharyngioma
Keywords: endoscopic endonasal surgery; pituitary adenoma; anti-fog device; suction irrigation; intracranial infection; randomized controlled trial
MeSH Terms: conditions — Pituitary Neoplasms; Craniopharyngioma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A single-use, sterile "anti-fog suction device" (a 4 Fr multi-channel silicone catheter) is introduced through the same nostril alongside the endoscope after induction of anaesthesia.
  The built-in micro-balloon is inflated with 1 ml air to anchor the tip in the posterior choana.
  Low-flow (2 L min-¹), filtered, room-temperature air is delivered through the central lumen, creating a gentle laminar stream that passes across the lens, continuously removing warm humid air and preventing condensation.
  Two side ports provide continuous low-pressure (-5 cmH₂O) suction of any blood or fluid, keeping the surgical field dry.
  The device remains in place for the entire operation and is removed before nasal packing. No extra incisions or sutures are required.
  Interventions: Device: Anti-fog suction device-a 4 Fr multi-channel silicone catheter
- Control group (No Intervention): Standard care: whenever the lens fogs, the scrub nurse withdraws the endoscope and irrigates its tip with 5-10 ml of 37 °C sterile saline from a 20 ml syringe. This manoeuvre is repeated as often as necessary (average 10-15 times per case).

INTERVENTIONS:
Device: Anti-fog suction device-a 4 Fr multi-channel silicone catheter — A single-use, sterile "anti-fog suction device" (a 4 Fr multi-channel silicone catheter) is introduced through the same nostril alongside the endoscope after induction of anaesthesia.
  The built-in micro-balloon is inflated with 1 ml air to anchor the tip in the posterior choana.
  Low-flow (2 L min-¹), filtered, room-temperature air is delivered through the central lumen, creating a gentle laminar stream that passes across the lens, continuously removing warm humid air and preventing condensation.
  Two side ports provide continuous low-pressure (-5 cmH₂O) suction of any blood or fluid, keeping the surgical field dry.
  The device remains in place for the entire operation and is removed before nasal packing. No extra incisions or sutures are required.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if the anti-fog suction device works to keep the surgical view clear during endoscopic nose-to-pituitary operations and whether it lowers the chance of brain-fluid infection. It will also learn about the safety of the device.

The main questions it aims to answer are:

* Does the device reduce the total time the surgeon has to stop because the lens fogs up?
* What medical problems (such as nose-bleed, tube blockage, or infection) do participants have when the device is used?

Researchers will compare the anti-fog device to the usual "water-squirt" method to see if the device works better.

Participants will:

* Have either the device or the usual water method applied during their planned pituitary surgery
* Stay in the hospital for the normal recovery period (about 3-5 days) and return for a routine check-up around day 7
* Allow the study team to record operating times, any fog-related pauses, and results of blood or spinal-fluid tests taken before and after surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Pre-operative MRI/CT diagnosis of pituitary adenoma or craniopharyngioma ≤ *3 cm without extensive skull-base invasion
* Scheduled for elective endoscopic endonasal transsphenoidal resection
* ASA physical status I-III
* Able and willing to give written informed consent and comply with follow-up

Exclusion Criteria:

* Severe nasal anatomical deformity, polyps, or prior nasal surgery preventing device placement
* Active nasal or systemic infection (WBC > 10 × 10⁹/L, CRP ≥ 10 mg/L)
* Known intracranial infection or ongoing CSF leak
* Coagulopathy (PT > 14 s or APTT > 45 s) or anticoagulation that cannot be stopped ≥ 7 days
* Allergy to silicone or medical-grade plastics
* Planned combined transcranial or transorbital approach
* Pregnancy or breastfeeding
* Psychiatric or cognitive disorder precluding informed consent or follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total duration of lens-fog interruptions (minutes) | Before the Nasal Packing(2 hours roughly)
  defined as the cumulative time from the moment the surgeon declares "lens fogged" until clear operative view is restored, measured with a stop-watch by the circulating nurse throughout the entire endoscopic endonasal procedure.

SECONDARY OUTCOMES:
post-operative intracranial infection rate | 7 days
  Incidence of post-operative intracranial infection within 7 days (positive CSF culture OR CSF WBC ≥ 10 × 10⁶/L with fever ≥ 38.5 °C).
Total irrigation fluid volume used intra-operatively (ml) | Before the nasal packing(2 hours roughly)
  Total irrigation fluid volume used intra-operatively (ml)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol